CLINICAL TRIAL: NCT01951898
Title: Effects of Montelukast on Airway Foxp3+ and CTLA4+CD25highCD4+ T Cells in Asthmatics
Brief Title: Effects of Montelukast on Airway Regulatory T Cells in Asthma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Tomotaka Kawayama, MD, Kurume University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KU-012012
Record Dates: First submitted 2012-05-02; First posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: asthma; regulatory T cells; leukotriene antagonist
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Montelukast (Active Comparator)
  Interventions: Drug: Montelukast
- Vitamin B6 (Sham Comparator)
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — 10mg/day, once a daily after dinner, for 28dyas

SUMMARY:
Montelukast is one of anti-inflammatory agents and a good controller for the patients with asthma. The hypothesis of the study is that the Montelukast will have airway anti-inflammatory effects and up-regulated regulatory T cells functions in asthma.

ELIGIBILITY:
Inclusion Criteria:

* asthma
* mild status
* stable status
* nonsmoker
* Positive of airway hyperresponsiveness (Methacholine-PC20<16mg/mL)

Exclusion Criteria:

* taken other asthmatic medications such as oral, injective, and inhaled steroids, leukotriene antagonists, oral, inhaled, and transdermal beta-agonists, theophylline, anti-histamine agents, anti-IgE antibodies and long acting muscarinic receptor antagonists.
* respiratory tract infections within 4wks
* moderate to severe other organ disorders
* active malignancies
* past histories of side effects of leukotriene antagonists
* psychological disorders
* pregnancy or nursing

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Montelukast will up-regulate airway regulatory T cell in the patients with asthma | 4wks of treatment period

SECONDARY OUTCOMES:
Montelukast will improve airway inflammation, lung function and hyperresponsiveness in the patients with asthma | 4wks of treatment periods

CONTACTS AND LOCATIONS:
Locations (1):
- Kurume University School of Medicine, Kurume, Japan